CLINICAL TRIAL: NCT04743232
Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) or COVID-19 Pandemic Resuscitation Plans and Decisions on Escalation and Limitation of Treatment
Brief Title: COVID-19 Resuscitation Plans and Decisions on Escalation and Limitation of Treatment
Acronym: CORDEAL
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the COVID pandemic became less severe (omikron)
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marc Schluep, Anesthesiologist-intensivist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NL76435
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Cardiac Arrest
MeSH Terms: conditions — COVID-19; Heart Arrest

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard practice (No Intervention): Standard practice concerning advanced care directives; care as usual
- Decision aid implementation (Experimental): Stepped-wedge implementation of the intervention
  Interventions: Other: Decision tool for clinicians

INTERVENTIONS:
Other: Decision tool for clinicians — Clinical decision aid, using a structured approach to advanced care directives and a comprehensive view of available risk scores.
  Arms: Decision aid implementation

SUMMARY:
During the Corona Virus Pandemic health care resources have become scare, and the pandemic has brought forth the need for risk stratification of patients suffering from COVID19 in order to allocate resources appropriately. One of scarcest resources is Intensive Care treatment, mostly related to the need for invasive ventilation or for (post) cardiac arrest care.

To identify patients for whom ICU-treatment is most successful and those for whom it would be futile, would allow for installing appropriate advanced care directives for escalation or limitation of treatment.

DETAILED DESCRIPTION:
Disease resulting from infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has a high mortality rate with deaths predominantly caused by respiratory failure. As of 1 September 2020, over 25 million people had confirmed coronavirus disease 2019 (COVID-19) worldwide and at least 850 000 people had died from the disease. As hospitals around the world are faced with an influx of patients with COVID-19, there is an urgent need for a pragmatic risk stratification tool that will allow the early identification of patients infected with SARS-CoV-2 who are at the highest risk of death to guide management and optimise resource allocation.

As is apparent not only from medical literature, but also from popular media, there is a need for risk stratification and decision aid. The problem with our current health care capacity mainly pertains to ICU-admissions. Ideally, clinicians would be able to predict who benefits from invasive ICU-treatment, and who does not. Subsequently, patients for whom ICU-admission is futile,doctors can install advanced care directives to refrain from escalation and limit the curative treatment they receive, and rather focus on palliation. As the investigators of this study previously discovered, patients are not unwilling to discuss these matters. In COVID-19 patients, three interventions seem logical to warrant special attention: ICU-admission, invasive ventilatory support and cardiopulmonary resuscitation. The latter because mortality in cardiac arrest patients with concurrent COVID appears higher than in non-COVID patients and performing CPR in patients with contagious diseases can potentially bring harm to health care providers.

Prognostic scores attempt to transform complex clinical pictures into tangible numerical values.

Dutch clinicians in general have been particularly busy identifying and providing prognostic scores for mortality and ICU-admission. Recent reviews listed many prognostic scores used for COVID-19, which varied in their setting, predicted outcome measure, and the clinical parameters included. It also highlights the importance of age, something that has been a subject to political debate. Therefore, in the past months, two Dutch research groups and one British group have developed two prognostic scores:

1. COVID Outcome Prediction in the Emergency department:

   COPE (ErasmusMC, NL)
2. Risk Stratification in the Emergency Department in Acutely Ill Older Patient:

RISE-UP (MUMC+, NL) 3. The International Severe Acute Respiratory and emerging Infections Consortium Coronavirus Clinical Characterisation Consortium of the World Health Organisation: 4C-score (UK)

In non-COVID patients, the Good Outcome for Attempted Resuscitation (GO-FAR) score serves as an acceptable prognostic tool for the prognosis of Cardiopulmonary Resuscitation (CPR). To date, no prognostic tool has been developed for CPR in COVID-patients. Last April, the Dutch board of intensive care medicine (NVIC) wrote a handbook to guide clinicians during the phase of the pandemic where resources would be limited to none (Code Black). In this handbook they summed up criteria in patients for whom ICU-admission would be futile or not-recommendable. Among these criteria was cardiac arrest. These criteria have however never been researched. Furthermore, although this handbook is necessary, there is no guidance for installing advanced care directives in the current stage of the pandemic, i.e. situations which are not Code Black - situations.

The aim of this study is to implement a clinical decision tool to aid clinicians in establishing advanced care directives about escalation and limitation of treatment in COVID-patients. The decision tool will provide two novelties: 1) A structured approach to discussing advanced care directives with patients who need to be admitted to hospital, and 2) A comprehensive oversight of available risk scores. The decision tool will not provide cut-off values or dichotomous decisions, this will be left to the discretion of the responsible physician. The secondary goal is to evaluate the use of this decision tool in terms of ICU-admissions, mortality and health care professionals' satisfaction with the implemented decision tool.

ELIGIBILITY:
Inclusion Criteria:

* adults with COVID19 (proven by polymerase chain reaction, or with strong clinical suspicion based on clinical features and/or radiodiagnostics)

Exclusion Criteria:

* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
ICU-admissions | before and after the intervention; total duration is 12 weeks.
  number of ICU-admissions at baseline and after implementation of the intervention

SECONDARY OUTCOMES:
Mortality | before and after the intervention; patient follow-up at 30 days and 1 year
  COVID mortality rates for hospital, ICU-mortality, 30-day and 1-year mortality.
Health care professionals' satisfaction | Measurements are repeated, before and after the intervention; total duration is 12 weeks.
  Health care professionals' satisfaction with the implemented decision tool and with the decision process as a whole. This will be measured via a structured questionnaire, using visual analogue scales (VAS, range 1-10) and Likert-scales for satisfaction scores.
Patient satisfaction | Measurement is only done once. In one group of patients before and another group after the intervention; total duration is 12 weeks.
  Patient satisfaction with the the communication in the hospital. This will be measured via a structured questionnaire, using visual analogue scales (VAS, range 1-10) and Likert-scales for satisfaction scores.

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - OLVG, Amsterdam, North Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Amsterdam UMC, Amsterdam
  - Rijnstate, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided